CLINICAL TRIAL: NCT03616743
Title: Effects of a Brief Pain and Smoking Cessation Intervention in Adults With Chronic Pain: A Randomized Controlled Trial
Brief Title: Brief Pain and Smoking Cessation Intervention in Adults With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, W. Michael Hooten, Professor of Anesthesiology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-000475
Record Dates: First submitted 2018-07-18; First posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-07

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief pain and smoking arm (Experimental): The experimental arm incorporated a novel psychoeducational component that addressed associations between cigarette smoking and chronic pain
  Interventions: Behavioral: Psychoeducation
- Brief smoking control arm (Active Comparator): The brief smoking control arm was comprised of the "5A's" of smoking cessation.
  Interventions: Behavioral: Brief smoking control arm

INTERVENTIONS:
Behavioral: Psychoeducation — Psychoeducation about the links between smoking and chronic pain.
  Arms: Brief pain and smoking arm
Behavioral: Brief smoking control arm — Psychoeducation about the general adverse effects of smoking.
  Arms: Brief smoking control arm

SUMMARY:
A brief smoking cessation intervention was developed to address smoking in the context of chronic pain to increase the intention to engage in smoking cessation treatment.

DETAILED DESCRIPTION:
The primary aim of this randomized controlled trial was to investigate the effects of a brief pain and smoking (BPS) cessation intervention on the willingness to consider quitting smoking in adults with chronic pain seeking treatment in a pain specialty outpatient clinic. The investigators hypothesized that participants randomized to the BPS intervention, relative to a brief non-tailored control smoking (BCS) intervention, would be more likely to self-report willingness to consider quitting smoking. Secondary aims included examining the effects of group allocation on the (1) interest in learning about smoking cessation programs; (2) willingness to consider scheduling a smoking cessation program; (3) scheduling a smoking cessation program; and (4) change scores of the Thoughts About Abstinence Scale (TAAS).

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* chronic pain of greater than 3 months duration
* smoke at least 10 cigarettes daily

Exclusion Criteria:

* cancer-related pain
* current participation in a smoking abstinence program
* current self-guided attempt to reduce or abstain from smoking
* use of other forms of tobacco including pipe, cigar or chew
* history of schizophrenia or other chronic psychotic disorder
* history of a dementing illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Self-report willingness to consider quitting smoking. | Immediate post-intervention assessment
  Single question with a binary self-report answer of Yes/No.

SECONDARY OUTCOMES:
Thoughts About Abstinence Scale | Pre-intervention and immediately post-intervention assessments
  The Thoughts About Abstinence Scale is a self-report questionnaire that assesses the desire to quit smoking, anticipated difficulty quitting, and anticipated success quitting smoking.

CONTACTS AND LOCATIONS:
Overall Officials: William M Hooten, MD, Principal Investigator — Professor of Anesthesiology

IPD SHARING:
Plan to Share IPD: No
Only a summary of group data will be shared.

REFERENCES:
- [Background] Hooten WM, Townsend CO, Hays JT, Ebnet KL, Gauvin TR, Gehin JM, Laures HJ, Patten CA, Warner DO. A cognitive behavioral smoking abstinence intervention for adults with chronic pain: a randomized controlled pilot trial. Addict Behav. 2014 Mar;39(3):593-9. doi: 10.1016/j.addbeh.2013.11.010. Epub 2013 Nov 21. PMID 24333035
- [Derived] Hooten WM, LaRowe LR, Zale EL, Ditre JW, Warner DO. Effects of a brief pain and smoking cessation intervention in adults with chronic pain: A randomized controlled trial. Addict Behav. 2019 May;92:173-179. doi: 10.1016/j.addbeh.2018.11.040. Epub 2018 Nov 28. PMID 30641335